CLINICAL TRIAL: NCT06663488
Title: Thoracic Spinal Versus Thoracic Epidural Anesthesia for Patients with Chronic Obstructive Pulmonary Disease Undergoing Supine Percutaneous Nephrolithotomy for Management of Renal Stones. a Prospective Double-blind Randomized Clinical Trial.
Brief Title: Thoracic Spinal Versus Thoracic Epidural Anesthesia for Patients with Chronic Obstructive Pulmonary Disease Undergoing Supine Percutaneous Nephrolithotomy for Management of Renal Stones.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Fouad Soliman, Principal investigator. Lecturer of Anesthesiology and ICU, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: 2011
Record Dates: First submitted 2024-10-18; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Postoperative Pain; Satisfaction with Care
Keywords: COPD; PNL; Thoracic epidural anesthesia; Thoracic spinal anesthesia
MeSH Terms: conditions — Pain, Postoperative; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Thoracic spinal anesthesia (Active Comparator): Thoracic spinal anesthesia: at T5-T6 or T6-T7 level with a 27G with 4 ml of isobaric bupivacaine 0.5% plus 0.5 ml of 250 ug morphine
  Interventions: Procedure: Thoracic spinal anesthesia
- thoracic epidural anesthesia (Active Comparator): Thoracic epidural anesthesia: The epidural needle was inserted At T6-8 space, After verification of the epidural space by resistance loss technique, a test dose of 2 ml of 0.5% bupivacaine will be injected. In the Cephalad direction, the epidural catheter was threaded 3 cm into the epidural space. A total dose of 8-12 ml 0.5 percent plain bupivacaine was injected
  Interventions: Procedure: Thoracic epidural anesthesia

INTERVENTIONS:
Procedure: Thoracic epidural anesthesia — The epidural needle was inserted At T6-8 space, After verification of the epidural space by resistance loss technique, a test dose of 2 ml of 0.5% bupivacaine was injected. In the Cephalad direction, the epidural catheter was threaded 3 cm into the epidural space. A total dose of 8-12 ml 0.5 percent plain bupivacaine was administered .
  Arms: thoracic epidural anesthesia
Procedure: Thoracic spinal anesthesia — Thoracic spinal anesthesia: At T5-T6 or T6-T7, a 27G needle was inserted. The needle's stylet will be removed and the hub observed for free flow of CSF; once flow of clear CSF, 4 ml of isobaric bupivacaine 0.5% plus 0.5 ml of 250 ug morphine was injected
  Arms: Thoracic spinal anesthesia

SUMMARY:
Owing to the elevated risk of perioperative comorbidities, chronic obstructive and restrictive pulmonary disorders can be a challenging task for the anesthetist. Endotracheal intubation and intermittent positive pressure ventilation (IPPV), two hallmarks of general anesthesia (GA), are known to increase the risk of serious complications such as barotrauma, laryngospasm, and bronchospasm. Patients who had neuraxial anesthesia had a lower rate of pulmonary and cardiac problems and deep venous thrombosis after surgery compared to those who received GA. Global Initiatives for Chronic Obstructive Lung Disease (GOLD) described COPD as a pulmonary disease with an inflammatory process that affects both the central and peripheral tracheobronchial tree, the pulmonary vasculature, and the pulmonary parenchyma. This persistent and cumulative process leads to the narrowing of the small airways, which is difficult to reverse, along with changes in the smooth muscle of the airway, increased secretion of mucus-secreting glands and goblet cells, and the development of perivascular pulmonary fibrosis. These changes contribute to the development of pulmonary hypertension and increase the workload on the right ventricle. Ultimately, COPD is characterized by the obstruction of airflow during expiration. When the small airway becomes inflamed, the condition is called "obstructive bronchiolitis," and when the lung tissue becomes destroyed, the condition is called "emphysema.". Impairment in ventilation and perfusion (V/Q) ratios and pulmonary mechanics come from air trapping and dynamic hyperinflation caused by obstruction in small airways.

Patients with COPD have a wide range of options for anesthesia, depending on illness stage, type of surgery, and length of operation. General anesthesia (GA) is known to increase the risk of problems for patients with COPD, especially when paired with endotracheal tube insertion and mechanical ventilation. Increased risk of hypoxemia and intra- and postoperative pulmonary complications; laryngospasm; bronchospasm; lung barotrauma; hemodynamic instability; hypercarbia; prolonged postoperative mechanical ventilation; and difficulty in weaning. To address these challenges, there has been a growing inclination towards employing various forms of regional anesthetic techniques whenever possible, including central neuraxial block. This approach aims to minimize the risks associated with general anesthesia and its potential complications, providing a safer alternative for COPD patients undergoing different types of surgical procedures. Regional blocking, as opposed to GA, has been found to improve pulmonary outcomes in patients with severe COPD and patients with normal lung function.

DETAILED DESCRIPTION:
The purpose of the current study is to identify, and evaluate the patient's outcome, and compare the use of either thoracic spinal anesthesia (TSA) or continuous thoracic epidural anesthesia (CTEA) as a single PNL anesthesia for stone kidney in patients with COPD.

Materials and methods:

After approval of the Scientific Research Ethical Committee, Faculty of Medicine, Sohag University, written informed consent will be taken from all patients.

Inclusion criteria:

- One hundred patients 45-80 years of age, with ASA physical status classes (II and III) complaining of COPD scheduled for various electives (PNL) for renal stone. All patients knew that they had COPD with stages I-III (mild to severe airflow limitation) with forced expiratory volume in 1 s (FEV1)/forced vital capacity (FVC) less than 70% of the normal value.

Exclusion criteria:

Patients reject neuraxial anesthesia and prefer GA. Local back infection. Lumbar or thoracic spine deformity. Coagulopathy or platelet dysfunction. Diabetic patients with peripheral or central neurological dysfunction. Pulmonary artery systolic pressure greater than 50 mmHg. Obesity (BMI >30). ASA physical status class less than III. PaCO2 of more than 45 mmHg and PaO2 of less than 60 mmHg on room air.

-Patients with allergy to local anesthetic (LA) drugs. On arrival at the operative room, a wide-bore peripheral intravenous line and a central line were inserted. Base level central venous pressure was recorded and then 500 ml lactated Ringer's solution was given. Arterial line penetration into the radial artery of the non-dependent arm for arterial blood gas (ABG) sampling and invasive blood pressure monitoring after ensuring a positive Allen test. ECG, pulse oximetry, noninvasive blood pressure, respiratory rate (RR), skin temperature, and the flow rate of urine were included in the monitoring.

Patients were randomly assigned into two equal groups, 50 patients in each.

First group: Thoracic spinal anesthesia (TSA group):

This group received segmental thoracic spinal anesthesia, first antiseptic preparation for cleaning the skin, then 1% lidocaine infiltrating the skin at the puncture site. Patients were put in a lateral decubitus or sitting position and puncture was performed via paramedian approach at the intersection of T5-T6 or T6-T7 in all patients with a 27G cutting needle (GMS). The needle's stylet was removed and the hub was observed for free flow of CSF; once the flow of clear CSF,4 ml of isobaric bupivacaine 0.5% plus 0.5 ml of 250 ug morphine was injected. The patient was then placed in the supine position.

The second group: Thoracic epidural anesthesia (TEA Group) The epidural needle will be as inserted At T6-8 space, After verification of the epidural space by resistance loss technique, a test dose of 2 ml of 0.5% bupivacaine was injected. In the Cephalad direction, the epidural catheter was threaded 3 cm into the epidural space. A total dose of 8-12 ml 0.5 percent plain bupivacaine was administered to the epidural catheter in 4 ml split aliquots at 5 min intervals after confirmation of catheter position. The bilateral sensory block in both midclavicular lines was tested every 2 minutes for loss of pinprick sensation. After 15 min, an additional 3-5 ml of bupivacaine was administered if the sensory block level was still below T5. Epidural anesthesia was retained when one-fourth to one-third of the initial LA dose was injected.

IF sensory regression occurred in two parts. For postoperative analgesia, epidural infusion of a mixture of 0.125 percent bupivacaine at a rate of 6-10 ml/h was maintained, with infusion rate adjustment according to VAS and side effects.

Oxygen was supplied to all patients by a nasal catheter at a rate of 2 L/min. Intraoperative hypotension [mean arterial pressure (MAP) <20% of preoperative value] was treated with intravenous 5 mg ephedrine in increments, Bradycardia [heart rate (HR) <55 beat/min] was treated with 0.5-2 mg intravenous atropine and the vomiting was treated by intravenous 10 mg metoclopramide. After surgery, all patients were transferred into the surgical PACU for monitoring, clinical evaluation, and management of any problem.

Supplemental epidural injections will be administered in aliquots of 5 ml isobaric bupivacaine 0.5% only if sensory block reseeds below the T5 dermatome, and systemic drugs cannot control the pain.

Intraoperative irritability was treated with re-assurance and midazolam bolus of 1-2 mg intravenously. Conversion to GA was done in cases where the surgeons faced a technical difficulty of the surgery or in case of lack of patient satisfaction with regional anesthesia at any time during the procedure.

Data that was recorded;

1. Patient's demographic data (age, body weight, sex ratio, ASA PS classes, duration of surgery, and blood loss).
2. Technical ease of the needle insertion and catheter threading through it. The degree of ease is classified as very easy, easy, difficult, and very difficult.
3. VAS score for pain as the postoperative analgesia was assessed by the VAS every 2 h.
4. Motor blockade was evaluated by the modified Bromage scale before starting the surgery, motor block at the end of the surgery, block regression in minutes (0 the patient can flex the extended leg at the hip, 1 can flex the knee but cannot flex the extended leg, 2 cannot move foot only, 3 cannot move foot).
5. Hemodynamic changes: HR and MAP, preoperatively (baseline values), intraoperatively every 5 minutes until the first 30 minutes then every 15 minutes until 4 hours, and postoperatively at 1 h after surgery,
6. Respiratory changes: RR (min), PaCO2 (mmHg), and PaO2 (mmHg) preoperatively (baseline values), intraoperatively at 30 min, 1 h, at end of surgery, and postoperatively at 1 h after surgery
7. The incidence of various side effects such as hypotension (MAP<20% of baseline value), bradycardia (HR<55 b/m), vomiting, pruritus, respiratory depression (RR<8 breath/min.
8. The patient was discharged from the postanesthetic care (PACU) after total regression of the block, provided that postoperative pain will be well controlled by systemic analgesics; in the form of ketolorac 30 mg IV, paracetamol 1 g IV, and/or nalbuphine 5-20 mg IM whenever needed. Epidural catheters were removed just prior to patients' discharge to their respective wards.
9. Patient and surgeon satisfaction was evaluated by using a four-point scale (4 is excellent, 3 is good, 2 is satisfactory, and 1 is poor), and the length of ICU stay. Pain severity was evaluated via VAS postoperatively at 2, 6, 12, and 24 h.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status classes (II and III) complaining of COPD scheduled for various elective (PNL) for renal stone.
* All patients known that they had COPD with stages I-III (mild to severe airflow limitation) with forced expiratory volume in 1 s (FEV1)/forced vital capacity (FVC) less than 70% of the normal value.

Exclusion criteria:

* Patients reject neuraxial anesthesia and prefer GA.
* Local back infection.
* Lumbar or thoracic spine deformity.
* Coagulopathy or platelet dysfunction.
* Diabetic patients with peripheral or central neurological dysfunction.
* Pulmonary artery systolic pressure greater than 50 mmHg.
* Obesity (BMI >30).
* ASA physical status class less than III.
* PaCO2 of more than 45 mmHg and PaO2 of less than 60 mmHg on room air.
* Patients with allergy to local anesthetic (LA) drugs.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-08-15 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-02 (Actual)

PRIMARY OUTCOMES:
1st analgesic requirment | 24 hours
  The time at which 1st analgesic was given
Respiratory monitoring | preoperatively (baseline values), intraoperatively at 30 min, 1 h, at end of surgery, and postoperatively at 1 h after surgery
  Respiratory rate (rate/min)

SECONDARY OUTCOMES:
PaCO2 | preoperatively (baseline values), intraoperatively at 30 min, 1 h, at end of surgery, and postoperatively at 1 h after surgery
  CO2 partial pressure (mmHg)
PaO2 | preoperatively (baseline values), intraoperatively at 30 min, 1 h, at end of surgery, and postoperatively at 1 h after surgery
  Oxygen partial pressure (mmHg)

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Sohag, Sohag Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No